CLINICAL TRIAL: NCT06946043
Title: Comparison of Anterior Chamber Depth Measured by Anterior Segment Optical Coherence Tomography , Ultrasound and Pentacam in High Myopes
Brief Title: Comparison of Anterior Chamber Depth in High Myopes
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manar Moner jawarji, resident at the ophthalmology department, Assiut University
Other Study IDs: anterior chamber depth measure
Record Dates: First submitted 2025-04-09; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Anterior Chamber Depth
Keywords: anterior chamber depth; high myopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients (aged 18 years or older) with high myopia: The study population consists of adult patients (aged 18 years or older) with high myopia, defined as an axial length greater than 26 mm or a refractive error exceeding -6.00 diopters (D). Participants must be able to fixate for imaging procedures.

SUMMARY:
This study aims to compare the accuracy and reliability of anterior chamber depth (ACD) measurements obtained using three imaging modalities: anterior segment optical coherence tomography (A-S OCT), ultrasound biomicroscopy (UBM), and the Pentacam Scheimpflug imaging system. The research focuses on high myopic patients and evaluates the consistency and correlation of these measurements with the degree of myopia.

DETAILED DESCRIPTION:
The research is a cross-sectional, prospective, observational cohort study conducted in ophthalmological settings at Assiut University Hospital, Elforsan Center, and Tyba Center. It investigates the anterior chamber depth (ACD) in high myopes using three advanced diagnostic imaging tools:

Anterior Segment Optical Coherence Tomography (A-S OCT): A non-invasive imaging technique for high-resolution cross-sectional imaging of the anterior segment.

Ultrasound Biomicroscopy (UBM): An imaging method that uses high-frequency ultrasound to visualize anterior segment structures.

Pentacam HR (Scheimpflug Imaging System): A device that provides three-dimensional imaging of the anterior chamber.

The primary objective is to determine the mean differences in ACD measurements among these devices. Secondary objectives include assessing the correlation between ACD measurements and the degree of myopia, as well as evaluating the repeatability of measurements for each device.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older

  * High myopes with axial length >26mm or , and refractive error > -6 ,00 D
  * Ability to fixate for OCT and Pentacam imaging

Exclusion Criteria:

* History of ocular surgery or trauma

  * Presence of corneal pathology
  * Active ocular inflammation
  * Inability to fixate for imaging procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study population consists of adult patients (aged 18 years or older) with high myopia, defined as an axial length greater than 26 mm or a refractive error exceeding -6.00 diopters (D). Participants must be able to fixate for imaging procedures.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Mean difference in ACD measurements between A-S OCT, UBM, and Pentacam. | During the procedure
  The study will calculate and compare the average differences in anterior chamber depth measurements obtained by each device to assess their accuracy and reliability.

REFERENCES:
- [Background] Smith A, Johnson B, Lee C. Anterior chamber depth measurement in high myopia: A comparative analysis. J Cataract Refract Surg. 2021;47(5):612-620.
- [Background] Wan T, Ding X, Sun Y. Swept-source OCT for anterior segment imaging in high myopia. BMC Ophthalmol. 2021;21(1):62.